CLINICAL TRIAL: NCT02341326
Title: Defective FGFR2 Signaling in the Small Airway Basal Progenitor Cells in COPD
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1311014509; R01HL123544 (NIH)
Record Dates: First submitted 2014-07-16; First posted 2015-01-19 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: COPD; Smoking; Lung Disorder
Keywords: Lung; COPD; smoking; Non-smoker
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — De-identified secondary lung tissue samples from deceased individuals (smokers or nonsmokers) with COPD or without COPD (normal lung donors without history of chronic lung disease) obtained via collaboration with Dr. Scott Randell, U North Carolina.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy nonsmokers: n=20 for Aim 1 n=20 for Aim 2
  Aim 1.To determine whether BC from the SAE of COPD smokers have reduced capacity to generate normally differentiated SAE, e.g initiate airway branching and repair in response to injury in vitro but generate airway epithelium with the phenotype similar to that present in SAE of COPD smokers in vivo.
  Aim 2.To test the hypothesis that FGFR2 signaling is necessary for normal SAE BC stem cell function and suppression of FGFR2 caused by inhibitors and smoking associated factors (EGF and TGF- beta)leads an altered stem cell functional phenotype similar to SAE BC from COPD smokers with reduced capacity as characterized by Aim 1.
- Healthy smokers: n=20- for Aim 1 n=20 for Aim 3
  Aim 1.To determine whether BC from the SAE of COPD smokers have reduced capacity to generate normally differentiated SAE, e.g initiate airway branching and repair in response to injury in vitro but generate airway epithelium with the phenotype similar to that present in SAE of COPD smokers in vivo.
  Aim 3.To assess the hypothesis that increasing FGFR2 signaling and suppressing smoking induced EGF receptors and TGF-beta pathways will restore the FGFR2 expression and normalize the capacity of SAE BC stem cells to generate and maintain normally differentiated SAE.
- COPD smokers: n=20- for Aim 1 n=20 for Aim 3
  Aim 1.To determine whether BC from the SAE of COPD smokers have reduced capacity to generate normally differentiated SAE, e.g initiate airway branching and repair in response to injury in vitro but generate airway epithelium with the phenotype similar to that present in SAE of COPD smokers in vivo.
  Aim 3.To assess the hypothesis that increasing FGFR2 signaling and suppressing smoking induced EGF receptors and TGF-beta pathways will restore the FGFR2 expression and normalize the capacity of SAE BC stem cells to generate and maintain normally differentiated SAE.

SUMMARY:
Early changes associated with the development of smoking-induced diseases, e.g., COPD and lung cancer (the two commonest causes of death in U.S.) are often characterized by abnormal airway epithelial differentiation. Airway basal cells (BC) are stem/progenitor cells necessary for generation of differentiated airway epithelium. Based on our preliminary observations on SAE BC cells and FGFR2 signaling, we hypothesized that suppression of FGFR2 signaling in the SAE BC stem/progenitor cells by cigarette smoking renders these cells less potent in generating and maintaining normally differentiated SAE, shifting these cells towards a COPD associated phenotype. To test this, SAE basal cells will be isolated from cultured cells obtained through bronchoscopic brushings and analyzed through in vitro assays for their stem/progenitor capacities.

DETAILED DESCRIPTION:
Changes within the small airways of the lungs represent the key element in the mechanism of COPD, as they precede the development of emphysema and contribute to the progressive decline in expiratory airflow. One of the key features of COPD is the remodeling of the small airway epithelium (SAE), and COPD SAE phenotypes are often induced by smoking and broad gene expression changes in the SAE. Many of the specific mechanisms for maintenance and regeneration of small airways and differentiated SAE in adult human lungs are largely unknown, but smoking associated defects in the maintenance of the SAE may be an early event of COPD. Preliminary data from murine studies have indicated that fibroblast growth factor receptor 2 (FGFR2) signaling is critical for lung architecture and development, and preliminary evidence has shown the FGFR2 pathway is down regulated within the small airway epithelium (SAE) of smokers and smokers with COPD. We hypothesize that the suppression of FGFR2 signaling in SAE BC stem cells by cigarette smoking causes these cells to become less potent, shifting the expression of normally differentiated SAE towards the COPD-associated small airway phenotype and therefore affecting the generation and maintenance of these cells. Using technologies established in our laboratories, pure populations of BC will be isolated from the SAE of healthy nonsmokers, healthy smokers, and COPD smokers. The stem/progenitor cell capacities of the SAE BC of each group will then be analyzed through the use of 3D modeling. The basic mechanisms of COPD will be tested by focusing on the phenotypes present in the lungs of COPD patients and comparison to their nonsmoker and healthy smoker counterparts. The 3 aims will be assessed in parallel, with all aims sharing in the biologic samples:

Aim 1 (n=60). To determine whether BC from the SAE of COPD smokers have reduced capacity to generate normally differentiated SAE, e.g initiate airway branching and repair in response to injury in vitro but generate airway epithelium with the phenotype similar to that present in SAE of COPD smokers in vivo.

Aim 2 (n=20). To test the hypothesis that FGFR2 signaling is necessary for normal SAE BC stem cell function and suppression of FGFR2 caused by inhibitors and smoking associated factors (EGF and TGF- beta) leads an altered stem cell functional phenotype similar to SAE BC from COPD smokers with reduced capacity as characterized by Aim 1.

Aim 3 (n=40). To assess the hypothesis that increasing FGFR2 signaling and suppressing smoking induced EGF receptors and TGF-beta pathways will restore the FGFR2 expression and normalize the capacity of SAE BC stem cells to generate and maintain normally differentiated SAE.

ELIGIBILITY:
Samples from newly recruited research subjects will be collected under the IRB approved protocol "Collection of Airway, Blood and/or Urine Specimens from Subjects for Research Studies" (IRB # 1204012331) or may have been collected under previous IRB approved collection protocols: #0005004439, #0005004440, and #0905010391.

Inclusion Criteria:

* Must be capable of providing informed consent
* Males and females, age 18 or older
* Nonsmoking, matched with other groups by age, sex, ethnic/racial group
* Good overall health without history of chronic lung disease, including asthma, and without recurrent or recent (within 3 months) acute pulmonary disease
* Normal physical examination
* Normal routine laboratory evaluation, including general hematologic studies, general serologic/ immunologic studies, general biochemical analyses, and urine analysis
* Negative HIV serology
* Normal chest X-ray (PA and lateral)
* Normal electrocardiogram
* Females - not pregnant
* No history of allergies to medications to be used in the bronchoscopy procedure
* Not taking any medications relevant to lung disease or having an effect on the airway epithelium
* Willingness to participate in the study

Exclusion Criteria:

* Unable to meet the inclusion criteria
* Pregnancy
* Current active infection or acute illness of any kind
* Current alcohol or drug abuse
* Evidence of malignancy within the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New York Metropolitan area residents
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

PRIMARY OUTCOMES:
Expression of FGFR2 and related pathways in SAE BC | 5 Years
  Measure of Expression of FGFR2 and related pathways in SAE BC

CONTACTS AND LOCATIONS:
Overall Officials: Renat Shaykhiev, MD, Principal Investigator — Weill Cornell Medical College, NY
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided